CLINICAL TRIAL: NCT00047866
Title: Brain Activation in Response to Motivational and Affective Stimuli: Pharmacological Manipulations
Brief Title: Brain Function in Response to Motivational Stimuli
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030013; 03-AA-0013
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-25

CONDITIONS: Drug Dependence
Keywords: Limbic System; Amphetamine; Dopamine; Brain Imaging; Cerebral Blood Flow; Cerebral Blood Volume; Alcoholism; Tyrosine Depletion; Amino Acids; Affect; Healthy Volunteer; HV
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

SUMMARY:
This study seeks more information about the biology of substance dependency by exploring the brain areas involved in feeling positive and negative emotions. Specifically, it will determine whether a brain chemical called dopamine affects activity in certain brain regions during performance of a game that involves winning and losing money. Brain activity will be examined using magnetic resonance imaging (MRI), a test that uses a magnetic field and radio waves to produce images of brain structure and function.

Young to middle-aged healthy adults may participate in this study. Candidates will be screened with a medical history, physical examination, electrocardiogram (EKG), psychiatric interview, and blood and urine tests. Participants will be assigned to one of the two study procedures, as follows:

Tyrosine/Phenylalanine

This study requires two overnight stays at the NIH Clinical Center. For each stay, subjects are admitted to the hospital the afternoon before the MRI scan. From the time of admission until after the scan, their diets are restricted to food relatively low in amino acids, prepared by NIH dietitians. The next day, participants undergo MRI scanning. For this procedure, the subject lies on a table that is moved into the scanner, a metal cylindrical machine. Earplugs are worn to muffle loud noises that occur with electrical switching of the radio frequency circuits. Imaging of brain structure takes about 10 to 15 minutes. Additional scans are then taken to measure brain activity while the subject plays simple computer games for money. These scans take about another 20 to 45 minutes. Five hours before the MRI, the subject drinks one of two beverages containing amino acids. A different beverage is given for each of the two visits: one drink lacks the essential amino acids tyrosine and phenylalanine, from which the body makes dopamine; the other contains balanced amounts of these two amino acids. Finally, subjects fill out mood-rating questionnaires before and after drinking each of the beverages.

Dextroamphetamine

This study requires two outpatient visits to the NIH Clinical Center. For one visit, participants are given an injection of 0.2 mg/kg body weight of the drug dextroamphetamine; for the other, they are given an injection of saline (salt water). After each injection, they undergo MRI scanning while playing computer games for money, as described above. They will fill out mood-rating questionnaires before and after each brain scan.

DETAILED DESCRIPTION:
The purpose of this protocol is to advance the understanding of the behavioral neurobiology underlying substance dependency by exploring regional brain activity in response to appetitive and aversive stimuli in human subjects. In this protocol, brain activation is the dependent measure, as measured by blood oxygenation level dependent (BOLD) signal acquired during functional magnetic resonance (fMRI) imaging. Previous work in this laboratory has found that cues of anticipated monetary reward versus threat of negative reinforcement causes increased BOLD signal in the nucleus accumbens (NAcc) and other parts of the ventral striatum. This protocol is intended to extend these findings by exploring whether the recently reported BOLD activation (a hemodynamic response) in certain brain regions in response to motivational cues can be perturbed by dopaminergic pharmacological manipulations.

In a series of two, repeated-measures, within-subject experiments, we propose to temporarily alter subjects' brain monoamine neurotransmitter systems with pharmacological interventions prior to presenting the subjects with appetitive and aversive visual stimuli as well as cues signaling potential punishment and reward. In the first experiment, brain catecholamine systems will be deactivated by dietary restrictions of amino acid precursors Tyrosine (Tyr) and Phenylalanine (Phe), respectively. In the second experiment, the brain dopamine (DA) release will be transiently increased with administration of dextroamphetamine (Amph). Based on a wealth of existent findings, we predict that acutely enhancing synaptic DA by Amph will augment reward-elicited activation in the ventral striatum. Conversely, acute dietary restriction of the DA precursor Tyr, (along with Tyr precursor Phe) will blunt this activation. Since substance use disorders (SUD) such as alcoholism may result from disordered neural systems regulating approach and avoidance behavior (with respect to the substance), this experiment can yield useful knowledge relevant to SUD.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Subjects are physically healthy as determined by medical evaluation at the NIAAA outpatient clinic. In particular, subjects must demonstrate no cardiovascular or blood pressure abnormalities, such as a resting blood pressure of 140/90 or greater. All values of laboratory test must be within the NIH defined normal range and all radiological and cardiac evaluations must be considered normal by the NIH radiologist or cardiologist reading the scan or record. As is usual clinical practice, in the case of minor abnormalities a lab test may be repeated to ensure the validity of the initial report.

Are between 18-65 years of age.

Have 20/20 vision or wear corrective contact lenses. Plastic glasses with pop-in lenses of different strengths are available in the NMR center for use with nearsighted subjects who do not wear contacts.

Have no ferromagnetic objects in their bodies which might be adversely affected by MRI (e.g. surgical clips; metal fragments in or near brain; eye or blood vessels; cardiac or neurological pacemaker; cochlear or eye implant - any doubt about absence of these objects will result in exclusion from this study).

Test HIV negative.

Have no indication of any organic brain syndrome.

Do not meet criteria for any present or past Axis I psychiatric disorder, including nicotine dependence. Smokers will be excluded.

Have no active homicidal or suicidal ideation, or active symptoms of post-traumatic stress disorder.

Are not currently receiving psychotropic medication or medication likely to affect brain neurotransmitter systems.

Have no indication of recent drug use as evidenced by urine drug screen and self-report.

Are not pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2002-10-12; Study Completion 2010-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Holland P, Mushinski M. Costs of alcohol and drug abuse in the United States, 1992. Alcohol/Drugs COI Study Team. Stat Bull Metrop Insur Co. 1999 Oct-Dec;80(4):2-9. PMID 10553265
- [Background] Koob GF. Neurobiology of addiction. Toward the development of new therapies. Ann N Y Acad Sci. 2000;909:170-85. doi: 10.1111/j.1749-6632.2000.tb06682.x. PMID 10911930
- [Background] Volkow ND, Wang GJ, Fowler JS, Logan J, Gatley SJ, Hitzemann R, Chen AD, Dewey SL, Pappas N. Decreased striatal dopaminergic responsiveness in detoxified cocaine-dependent subjects. Nature. 1997 Apr 24;386(6627):830-3. doi: 10.1038/386830a0. PMID 9126741